CLINICAL TRIAL: NCT06074796
Title: The Determinants of Fertility Preservation in TRANSgender Patients (FP-TRANS).
Brief Title: The Determinants of Fertility Preservation in TRANSgender Patients.
Acronym: FP-TRANS
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mikael AGOPIANTZ, head of the ART center, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI127-413
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Fertility Preservation; Transgender; Transgenderism
Keywords: transgender; fertility preservation; parenthood; social determinants
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender patients: Patients included are transgender patients who have had routine consultations as part of the transition process for transgender patients, done in the reproductive medicine department of the regional university hospital centre in Nancy. Exclusion criteria : minors, patients under guardianship or trusteeship.
  French laws allow embryo transfer until 45 years for women and sperm reuse up to 60 years for men, so patients older have been excluded.
  Interventions: Behavioral: No intervention.

INTERVENTIONS:
Behavioral: No intervention. — No intervention. This is a retrospective study. Data will have been collected in routine consultations as part of the transition process for transgender patients.
  Description of the collected informations : gender of destination, BMI, siblings, children, moral, previous hormone therapy, when the project was born, change of marital status desired or carried out, ALD status, psychiatric assessment, desire for future care for the transition course. Desire to preserve erectile function, parenthood desire, couple projections, type of couple, cryopreservation desired, done or not, desire of pregnancy, ultrasound count of antral follicles, initial hormone assays and tests : BMD, pelvic ultrasound? Data relating to stimulation and ovarian puncture and sperm collection.

SUMMARY:
The study is monocentric, retrospective, non-interventional and does not involve human subjects.

The main objective is to compare the profiles of transgender patients who undergo fertility preservation with those who do not.

The secondary objectives are to define the rate of recourse to fertility preservation, determine the proportion of patients wishing to become parents.

Statistical analysis will be carried out with a view to highlighting significant determinants in transgender patients by comparing those who undergo fertility preservation with those who do not.

The data will have been collected during routine consultations as part of the transition process for transgender patients. This is taking place in the reproductive medicine department of the regional university hospital centre in Nancy.

DETAILED DESCRIPTION:
This study aims to assess the determinants of fertility preservation (FP) among transgender patients at the University Regional Hospital Center (CHRU) of Nancy. The secondary objective was to establish a database to gain a deeper understanding of the challenges related to fertility preservation in the context of a transition project and thus provide more tailored support to transgender patients.

The primary endpoint is the significativity of profiles elements of transgender patients who undergo fertility preservation with those who do not.

It may help the understanding of the determinants of fertility preservation in transgender patients.

We expect to include between 200 and 300 patients. The data will be transcribed onto the anonymised data collection Excel sheet. Statistical analysis of qualitative and quantitative data will be carried out with a view to highlighting significant determinants in transgender patients by comparing those who undergo fertility preservation with those who do not.

The study is monocentric, retrospective, non-interventional and does not involve human subjects. In fact, this research is based on existing data, extracted from patient files in the médifirst software. The data will have been collected during routine consultations as part of the transition process for transgender patients. This is taking place in the reproductive medicine department of the regional university hospital centre in Nancy.

ELIGIBILITY:
Inclusion Criteria:

* Transgender patients who consulted the Assisted Reproductive Technology centre of the Nancy Regional University Hospital, between 1st January 2020 and 30th June 2023. The consultations occurred for the start of transition care, for follow-up or for a parenting project for transgender patients.

Exclusion Criteria:

* minors
* patients under guardianship or under tutelage

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — transgender patients
Study Population: Adult transgender patients who consulted the Assisted Reproductive Technology centre of the Nancy Regional University Hospital, between 1st January 2020 and 30th June 2023. The consultations occurred for the start of transition care, for follow-up or for a parenting project for transgender patients.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
significant result p < 0.05 of qualitative and quantitative data | Statistiques Will be done by December 2023.
  The significance of statistical tests (significant result p < 0.05) will show whether or not there are emerging determinants in each of the 2 groups: fertility preservation done / not done. Qualitative data will be available in the medical files created during the appointments of transgender patients who have consulted the Reproductive Medicine Department.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael AGOPIANTZ, PHD MCU, Principal Investigator — CentralHNF Nancy Regional University Hospital
Locations (1):
- Centre AMP Maternité Régionale de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mattelin E, Strandell A, Bryman I. Fertility preservation and fertility treatment in transgender adolescents and adults in a Swedish region, 2013-2018. Hum Reprod Open. 2022 Feb 21;2022(2):hoac008. doi: 10.1093/hropen/hoac008. eCollection 2022. PMID 35309678